CLINICAL TRIAL: NCT00972387
Title: "Nutritional Ergogenic Aids: The Effects of Carbohydrate-Protein Supplementation During Endurance Exercise"
Brief Title: Carbohydrate-Protein Supplementation During Endurance Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: University of TN IRB 7959-B
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Supplementation During Endurance Performance
Keywords: carbohydrate-protein; endurance exercise; supplement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Order 1 (Active Comparator): Supplement order for each time trial run, 1-4 respectively: CHO, CHO-P, CHO-CHO, PLA
  Interventions: Dietary Supplement: CHO, CHO-P, CHO-CHO, PLA
- Order 2 (Active Comparator): Supplement order for each time trial run, 1-4 respectively: CHO-P, CHO-CHO, PLA, CHO
  Interventions: Dietary Supplement: CHO-P, CHO-CHO, PLA, CHO
- Order 3 (Active Comparator): Supplement order for each time trial run, 1-4 respectively: CHO-CHO, PLA, CHO, CHO-P
  Interventions: Dietary Supplement: CHO-CHO, PLA, CHO, CHO-P
- Order 4 (Active Comparator): Supplement order for each time trial run, 1-4 respectively: PLA, CHO, CHO-P, CHO-CHO
  Interventions: Dietary Supplement: PLA, CHO, CHO-P, CHO-CHO

INTERVENTIONS:
Dietary Supplement: CHO, CHO-P, CHO-CHO, PLA — The CHO supplement will be administered during trial 1. The CHO-P will be administered during trial 2. The CHO-CHO supplement will be administered during trial 3. The PLA supplement will be administered during trial 4. This is the order of supplement administration for subjects randomly assigned to this order group.
  Arms: Order 1
Dietary Supplement: CHO-P, CHO-CHO, PLA, CHO — The CHO-P supplement will be administered during trial 1. The CHO-CHO will be administered during trial 2. The PLA supplement will be administered during trial 3. The CHO supplement will be administered during trial 4. This is the order of supplement administration for subjects randomly assigned to this order group.
  Arms: Order 2
Dietary Supplement: CHO-CHO, PLA, CHO, CHO-P — The CHO-CHO supplement will be administered during trial 1. The PLA will be administered during trial 2. The CHO supplement will be administered during trial 3. The CHO-P supplement will be administered during trial 4. This is the order of supplement administration for subjects randomly assigned to this order group.
  Arms: Order 3
Dietary Supplement: PLA, CHO, CHO-P, CHO-CHO — The PLA supplement will be administered during trial 1. The CHO will be administered during trial 2. The CHO-P supplement will be administered during trial 3. The CHO-CHO supplement will be administered during trial 4. This is the order of supplement administration for subjects randomly assigned to this order group.
  Arms: Order 4

SUMMARY:
The purpose of this study is to assess whether the greater performance benefits from ingesting carbohydrate-protein supplements during endurance running, in comparison to the traditionally used carbohydrate supplement, is attributed to the extra calories contained in the carbohydrate-protein supplement or the presence of protein.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the performance benefits from consuming a carbohydrate-protein (CHO-P) supplement, such as Accelerade, during endurance exercise, as opposed to the traditionally used carbohydrate (CHO) supplement, such as Gatorade, are attributed to the extra calories in the CHO-P supplement or the presence of protein alone in comparison to CHO supplements. Numerous studies comparing CHO and CHO-P supplements on endurance performance have found contradicting results in terms of CHO-P supplementation and performance benefits. While physiological mechanisms have been proposed as to why the CHO-P supplements elicit greater performance, research has yet to determine why some studies have found this, especially while other studies have found no performance benefits from CHO-P supplementation. This inconsistency in research may be due to the caloric difference between supplements tested; due to the addition of protein, the CHO-P supplement contains more calories per serving than the CHO supplement. As a result, this study will be comparing 4 different supplements during endurance exercise, a CHO-P supplement, CHO supplement, a double carbohydrate supplement (CHO-CHO), and a placebo (PLA). The CHO and CHO-P supplement will be matched for CHO content, whereas the CHO-P and CHO-CHO supplements will be matched for total caloric content. Participants will be asked to run four 12-mile runs on 4 separate occasions, approximately 7-10 days apart, and will be blinded to supplement content and order of supplement administration among trials. The 12-mile run will elicit an exercise bout greater than 60 minutes, which is relevant when supplementing exercise with CHO or CHO-P. Performance will be assessed via time it takes to complete both the 12-mile run and the 1.6 mile maximal effort at the end of the run.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-55 years old
* BMI in the healthy range, 18.5-24.9
* Run 45-90+ minutes at least 4 days per week
* Engage in running this frequency and duration for at least 4 weeks prior to the phone screen
* Engage in a run consisting ≥10 miles in length for at least 2-4 occasions per month for at least 2 months prior to the phone screen
* No previous history of heart conditions
* No shortness of breath or chest pain experienced during running or daily activities
* No bone or joint problems experienced during running or daily activities

Exclusion Criteria:

* Females and males under the age of 18 and over the age of 55
* Females are excluded from this study in order to prevent any potential factors associated with the female athlete triad and endurance performance outcomes.
* BMI below 18.5 or greater than 24.9
* Does not meet all other criteria listed (#3-6)
* Allergies to products containing milk, soy, or aspartame
* Severe allergies to eggs, wheat, tree nuts, fish, crustaceans, shellfish products (Accelerade, the CHO-P supplement, is made in a facility that processed these products)
* Refusal to consume any of the supplements, and/or extreme dislike of the supplements
* Refusal to complete the specified distance of the time trials

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time it takes to complete each 12-mile time trial run | 4 days
Time it takes to complete the 1.6 mile maximal effort at the end of the 12 mile run. | 4 days

SECONDARY OUTCOMES:
Heart Rate at the beginning of each time trial, start of the maximal effort, end of the run. | 4 days
Rating of perceived exertion through out the duration of the 12 mile time trial run. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Study Chair — University of Tennessee, Knoxville
Locations (1):
- Health Physical Education and Recreation Building, Knoxville, Tennessee, United States

REFERENCES:
- See also: Related Info — http://nutrition.utk.edu/healthy-eating-and-activity-laboratory/